CLINICAL TRIAL: NCT05481632
Title: Validating the Safety and Effectiveness of ENDOANGEL Lower Gastrointestinal Endoscope Image Auxiliary Diagnostic Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Wuhan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EndoAngel -CTP-01
Record Dates: First submitted 2022-07-22; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Intestinal Polyps
MeSH Terms: conditions — Intestinal Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician AI-assisted diagnosis group (Experimental)
  Interventions: Other: Endoangel assisted the process of colonoscopy
- Physician Independent Diagnostic Group (Sham Comparator)
  Interventions: Other: Colonoscopy was performed without endoangel assistance

INTERVENTIONS:
Other: Endoangel assisted the process of colonoscopy — Endoangel assisted doctors to detect polyps
  Arms: Physician AI-assisted diagnosis group
Other: Colonoscopy was performed without endoangel assistance — Polyps were detected without ENDOANGEL assistance
  Arms: Physician Independent Diagnostic Group

SUMMARY:
To evaluate the safety and effectiveness of ENDOANGEL Lower Gastrointestinal Endoscope Image Auxiliary Diagnostic Software developed and manufactured by Wuhan ENDOANGEL Medical Technology Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 75 years old, male or female;
* Subjects with colonoscopy diagnosis and screening needs;
* Sign the Written Informed Consent Form;
* With full capacity for civil conduct.

Exclusion Criteria:

* History of acute myocardial infarction (within 6 months), severe heart, liver, and renal insufficiency or mental disease;
* Patients who are taking aspirin, warfarin, and other anticoagulants;
* Patients with inflammatory bowel disease, or polyposis syndromes, or confirmed or highly suspected colon cancer;
* History of colorectal surgery;
* Patients with familial adenomatous polyposis;
* Pregnant women (if the subject is a woman of reproductive age and cannot confirm whether she is pregnant, a pregnancy test is required);
* Patients who are participating in clinical trials of other drugs or medical devices;
* Patients who are not eligible to participate in this clinical trial in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
sensitivity of polyps identification | 3 months
  The numerator is the number of true positives and the denominator is the total number of true positives and false negatives.
specificity of polyps identification | 3 months
  The numerator is the number of true negatives and the denominator is the total number of true negatives and false positives.

SECONDARY OUTCOMES:
Polyp detection rate | 3 months
  The numerator is subjects with polyps detected and the denominator is all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China